CLINICAL TRIAL: NCT05425914
Title: Impact of Vitamin D3 Supplementation in Non-Sjogren Dry Eye Patients With Low Serum Vitamin D Level
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Bushra Kanwal, Principal Investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUF Faisalabad
Record Dates: First submitted 2022-06-11; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Dry Eye Syndromes; Hypovitaminosis D
Keywords: Artificial tears.; Dry eye syndrome.; vitamin d deficiency.
MeSH Terms: conditions — Dry Eye Syndromes; Vitamin D Deficiency | interventions — Vitamin D; Lubricant Eye Drops

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment (Active Comparator): Receiving conventional dry eye treatment in the form of artificial tears four times per days for 90 days.
  Interventions: Drug: Artificial tear
- Vitamin D3 Supplementation (Experimental): Receiving vitamin d3 supplementation 6000IU per day along with artificial tears for 90 days.
  Interventions: Drug: Vitamin D; Drug: Artificial tear

INTERVENTIONS:
Drug: Vitamin D — New treatment option for dry eye patients with low serum vitamin D Level
  Arms: Vitamin D3 Supplementation
Drug: Artificial tear — Conventional dry eye treatment

SUMMARY:
Dry eye disease is multifactorial, ocular inflammatory condition causing irritation, stinging sensation, uneasiness and blurring. Non-Sjogren syndrome occurs due to absent or dysfunction of lacrimal gland. Fat soluble vitamin D act as an agent against inflammation and its deficiency may result in various inflammatory diseases including dry eye. Purpose of this study is evaluation of vitamin D3 supplementation role in treating non-Sjogren dry eye along with conventional treatment by using artificial tears in patients with hypovitaminosis D. A prospective study was conducted in Rural health center(RHC) Buchal Kalan on 108 patients presenting with non-Sjogren dry eyes and low serum vitamin D levels. Patients were subjected to the following examination; best corrected visual acuity (BCVA), slit-lamp examination, applanation tonometry, fundoscopy, tear breakup time (TBUT) after fluorescein staining, Schirmer tear test, numerical pain rating scale (NPRS) and ocular surface disease index (OSDI) score on day 0, 15, 30, 60 and 90. Vitamin D levels was assessed by electrochemiluminescence immunoassay (ECLIA) based analyzer. The sample was randomly divided into two groups by non-probability purposive sampling. Group 1 received only artificial tears 4times/day while group 2 were given oral vitamin D3 supplementation of 6000 international unit (IU) daily along with artificial tears. Impact of oral vitamin D3 supplementation on non-Sjogren dry eyes was assessed by comparing means of ocular parameters of both groups over different period of time by using Mann-Whitney Test and Friedman Test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-Sjogren dry eyes with low serum vitamin D level.
* Both gender.
* Age group will be 20-50 years of age.
* Cooperative patients.

Exclusion Criteria:

* Autoimmune diseases (such as Sjogren syndrome and lupus syndrome).
* All ocular pathologies except dry eyes.
* All systemic pathologies that affects tear layers.
* All non- cooperative patients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Tear Breakup time in seconds | 90 days
  Improvement after vitamin D3 supplementation over a period of time
Schirmer test score in millimeters | 90 days
  Improvement after vitamin D3 supplementation over a period of time

SECONDARY OUTCOMES:
Ocular surface disease index score in units | 90 days
  Change in both groups after treatment. Values ranges from 0 to 100. Higher score indicates worse condition.
Numerical Pain Rating Scale | 90 days
  Change in both groups after treatment. Values ranges from 0 to 10 wher 0 indicates no pain while 10 indicates worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Kanwal, MPO, Principal Investigator — The University of Faisalabad
Locations (1):
- RHC Buchal Kalan, Chakwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Plan to share results only due to confidentiality